CLINICAL TRIAL: NCT06469983
Title: Multicentric Study on Combined Verticalization and Mobilization in Patients With Severe Acquired Brain Injury: A Randomized Controlled Trial
Brief Title: Robotic vs. Traditional Verticalization in Patients With Severe Acquired Brain Injury: a Randomized Controlled Trial
Acronym: VEM-sABI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Estraneo (Other)
Collaborators: Istituti Clinici Scientifici Maugeri SpA (Other); Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor-Investigator, Anna Estraneo, Senior Researcher, Fondazione Don Carlo Gnocchi Onlus
Organization: Fondazione Don Carlo Gnocchi Onlus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VEM-sABI
Record Dates: First submitted 2024-06-14; First posted 2024-06-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acquired Brain Injury; Disorder of Consciousness
Keywords: Disorders of Consciousness; rehabilitation; verticalization; robotic
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Double blind could not be applicable since a physical therapist could be blinded due to the nature of the intervention (VEM or SV). However, clinical evaluation will be performed by an examiner blind to the patient' group of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Verticalization (Experimental): Erigo® gradual verticalization (from supine position up to maximum 90°, in 3 steps), depending on the patient's vital signs compliance. The Erigo verticalization is coupled with the rhythmic passive movement of the lower limbs ensuring the more normal range of motion (ROM) and the alternation of loading and unloading of the lower limbs, based on patient's osteo-articular condition (e.g., ROM=45°; cadence=min. 24 steps per minute).
  Interventions: Device: ErigoBasic or ErigoPro®
- Traditional Verticalization (Active Comparator): gradual verticalization (from supine position up to maximum 90°, in 3 steps), depending on the patient's vital signs compliance, using a traditional standing device (i.e., non-robotic traditional tilt table)
  Interventions: Behavioral: Traditional Verticalization

INTERVENTIONS:
Device: ErigoBasic or ErigoPro® — Static bed with integrated robotic stepper (ErigoBasic) and optionally integrated with Functional Electrical Stimulation (FES ErigoPro®). The Erigo is a robot designed to be used for early functional mobilisation of patients with neurological manifestations or who are bedridden, even in intensive care. It is a tilt table equipped with an integrated passive stepper controlled by microprocessors that generate physiological leg movements: the patient's thighs are secured by straps to the movement mechanisms and the feet are secured to plates equipped with shock absorbers, while the upper body is held in place by a sling integrated into the table. Erigo provides active functions: gradual elevation in orthostatism up to 90°, controlled and independent mobilisation of the lower limbs, and functional stimulation.
  Arms: Robotic Verticalization
Behavioral: Traditional Verticalization — gradual verticalization (from supine position up to maximum 90°, in 3 steps), depending on the patient's vital signs compliance, using a traditional standing device (i.e., non-robotic traditional tilt table)
  Arms: Traditional Verticalization

SUMMARY:
In the rehabilitation project for patients with severe Acquired Brain Injury (sABI), it is essential to include exercises that facilitate the recovery of the upright position (or verticalization). Recently, tilt-table equipped with the robot-assisted lower limbs cyclic mobilization has been proposed as a safe and suitable device for accelerating the adaptation to vertical posture in bedridden patients with brain-injury since the acute phase. The present multicentre study aims at evaluating the effectiveness of robotic assisted verticalization plus mobilization (VEM) versus traditional verticalization (TV) in a large cohort of patients with sABI.

DETAILED DESCRIPTION:
Background Italian Consensus on rehabilitation of patients with severe acquired brain injury (sABI) and recent American Academy of Neurology guidelines on patients with sABI and prolonged disorder of consciousness (pDoC) provided recommendations for admission of such complex disabled patients to inpatient specialized rehabilitation units with high expertise on multidisciplinary care.

In such dedicated settings (in Italy named as high specialty rehabilitation for sABI, Cod 75) a comprehensive standard rehabilitation programme includes positioning, prolonged passive range of motion exercises, and splinting protocols to prevent or remediate neuromuscular complications (contractures, spasticity, and heterotopic ossifications). Simultaneously, basic multi-sensory stimulation or targeted cognitive training should be implemented for facilitating cognitive functioning recovery. In the rehabilitation project for patients with sABI, it is essential to include exercises that facilitate the recovery of the upright position (or verticalization), in order to prevent secondary complications from immobility (e.g., stasis pneumonias, deep vein thrombosis), to facilitate the stabilization of the haemodynamic balance (known to be altered in this population after the acute event), to promote the improvement of cognitive performance (especially vigilance and attention), and to improve the muscular-cutaneous trophism. Verticalization with traditional tilt-table training can show several adverse events: no leg movements during tilt-table verticalization lead to limited musculoskeletal and cardiovascular response; 2. pooling of blood in the lower extremities which can lead to a drop of the central blood and hypotension; 3. It requires substantial modification of cardiovascular therapy due to presyncope symptoms.

More recently, tilt-table equipped with the robot-assisted lower limbs cyclic mobilization has been proposed as a safe and suitable device for accelerating the adaptation to vertical posture in bedridden patients with brain-injury since the acute phase. However, contrasting, and inconclusive effects of controlled verticalization on functionality, gait/balance and level of consciousness in patients with sABI have been found, likely because of the limited methodological quality of the available clinical trials. All studies present some concerns such as small cohorts or heterogeneous cohorts of patients with sABI (e.g., chronic patients with sequelae of sABI) or the randomization process is not described.

The present multicentre study aims at overcoming these limitations evaluating the effectiveness of robotic assisted verticalization versus traditional verticalization (TV) in a large cohort of patients with sABI. Standardized and validated clinical tools will be used for evaluating effect on patient's motor, cognitive and functional performances. Additional markers will be used as outcome measures for investigating possible brain plasticity. Neurophysiological findings (e.g., EEG background activity and reactivity and quantitative EEG metrics) and blood biomarkers have been correlated to cognitive performance and assist prognostication in patients with sABI and pDoC34,. Brain-derived neurotrophic factor, BDNF, a neurotrophin involved in neurogenesis and synaptic plasticity can be upregulated by physical exercise. However, a recent study showed that BDNF serum levels do not change after robotic assisted verticalization in patients with pDoC. Neurofilament light chain, NF-L, a marker of primary and secondary neurodegeneration in sABI was linked to long-term axonal degeneration and poor outcome. Glial fibrillary acid protein, GFAP, a filament protein is related to brain function recovery.

Methods 118 patients will be randomized to receive either VEM or TV at the same period of the day throughout the experiment. In the week before starting study protocol, the VEM and TV groups will undergo a preliminary "tolerance session test" of gradual verticalization (starting from 10 min and then progression toward 30 min).

The study protocol will involve 5 VEM or 5 TV sessions per week for 4 weeks (total 20 sessions). Each daily VEM or SR session last 30 minutes.

VEM protocol and parameters: Erigo® gradual verticalization (from supine position up to maximum 90°, in 3 steps), depending on the patient's vital signs compliance. The Erigo verticalization is coupled with the rhythmic passive movement of the lower limbs ensuring the more normal range of motion (ROM) and the alternation of loading and unloading of the lower limbs, based on patient's osteo-articular condition (e.g., ROM=45°; cadence=min. 24 steps per minute).

TV protocol: consists in gradual verticalization (from supine position up to maximum 90°, in 3 steps), depending on the patient's vital signs compliance, using a traditional standing device (i.e., non-robotic traditional tilt table) Both groups received an additional 60 minute-comprehensive daily (60 minutes) rehabilitation programme in the 3 months of the study. This programme consists of alternate bed positioning, passive limbs mobilization, activities to increase arousal (e.g., multisensory stimulation), language and swallowing therapy based on patient's functional condition.

Primary endpoint Level of Cognitive Functioning, LCF Secondary endpoints Modified Ashworth scale, MAS; Muscle Research Council, MRC (EpDoC) pDoC reflex movement to nociceptive stimulation (pDoC); Disability Rating Scale, DRS; Adverse Events Report (AER)+Agitation Behavior Scale and Nociception Coma Scale respectively; System Usability Scale (SUS); modified Barthel Index (mBI).

Exploratory endpoints Coma Recovery-Scale Revised, CRS-R (in pDoC) EEG architecture (e.g., microstates, functional connectivity, and complexity measures) Blood biomarkers (i.e., BDNF, NF-L, and GFAP); Fondazione Don Gnocchi-Clinical Complications Scale, FDG-CCS.

Adverse Events Report (weekly from enrolment through termination of RV or TV protocol). During VEM session Heart rate (HR), mean arterial pressure (MAP), oxygen saturation (SaO2), agitation, and pain will be monitored. Additionally, agitation and pain will be measured by the Agitation Behavior Scale and Nociception Coma Scale respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* sABI due to traumatic, vascular, anoxic, or mixed etiology;
* Stable behavioral/cognitive diagnosis on at least 4 behavioral evaluations in 1 week using the Italian version of the CRS-R in patients with pDoC, or the LCF-based cognitive assessment in patients with eDoC;
* Time post-injury between 28 days and 6 months [1];
* Not recovered upright station;
* Written informed consent by the patient's legal rep-resentative/primary caregiver.

Exclusion Criteria:

* Severe medical conditions hampering verticalization (e.g., severe hypotension or conditions realizing hemodynamic instability, end stage or severe symptomatic heart failure with reduced ejection fraction, cardiac arrhythmia of new diagnosis or arrhythmic flare, severe hepatic failure, chronic severe lower limb arterio-venous disease, sep-sis/septic shock, thrombus venous embolism of new diag-nosis, severe autonomic dysreflexia);
* Severe medical conditions hampering lower limb mobili-zation (e.g., fractures, heterotopic ossifications);
* Severe medical conditions impacting EEG activity (e.g., sub-continuous or abundant EEG epileptiform abnormali-ties);
* Severe medical conditions influencing conscious-ness/cognitive status, such as severe hyponatremia or hy-poglycemia;
* Contraindications to the use of Erigo®Basic and/or Eri-go®Pro (Hocoma, Volketswil, Switzerland) as per technical data sheet (see Appendix A);
* Presence of prohibited drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Levels of cognitive functioning | 5 weeks
  A clinical scale assessing global cognitive functioning in patients emerged from a disorder of consciousness. Higher scores indicate a higher cognitive functioning

SECONDARY OUTCOMES:
Modified Ashworth scale | 5 weeks - 1 month after treatment
  A clinical scale assessing spasticity. Higher scores indicate a more severe spasticity
Medical Research Council Scale | 5 weeks - 1 month after treatment
  A clinical scale assessing muscle functioning. Higher scores indicating a better functioning
modified Barthel Index | 5 weeks - 1 month after treatment
  It is a measure of functional disability, with higher scores indicating higher functional independence
Disability Rating Scale | 5 weeks - 1 month after treatment
  It is a measure of functional disability, with higher scores indicating higher disability
System Usability Scale | 5 weeks - 1 month after treatment
  It is a measure of usability and compliance. Higher scores indicate a better performance

OTHER OUTCOMES:
Spectral metrics | 5 weeks - 1 month after treatment
  Measure of quantitative EEG. Higher values indicate a better functional connectivity
Microstate metrics | 5 weeks - 1 month after treatment
  Measure of quantitative EEG. Higher values indicate a better functional connectivity
Connectivity metrics | 5 weeks - 1 month after treatment
  Measure of quantitative EEG. Higher values indicate a better functional connectivity
Brain-derived neurotrophic factor | 5 weeks - 1 month after treatment
  Blood biomarker. Higher value indicate higher brain plasticity
Neurofilament-Light | 5 weeks - 1 month after treatment
  Blood biomarker. Higher value indicate higher brain plasticity
Glial fibrillary acidic protein | 5 weeks - 1 month after treatment
  Blood biomarker. Higher value indicate higher brain plasticity
Fondazione Don Gnocchi-Clinical Complications Scale | 5 weeks - 1 month after treatment
  A clinical scale assessing clinical complications. Higher scores indicate more and more severe clinical complications
Coma Recovery Scale-Revised total score | 5 weeks - 1 month after treatment
  A clinical scale assessing the level of consciousness in patients with disorders of consciousness. Higher scores indicate a higher level of consciousness
Levels of cognitive functioning | 1 month after treatment
  A clinical scale assessing global cognitive functioning in patients emerged from a disorder of consciousness. Higher scores indicate a higher cognitive functioning

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Polo Specialistico Riabilitativo Fondazione Don Carlo Gnocchi ONLUS, Sant'Angelo dei Lombardi, Avellino
  - IRCCS Maugeri Telese Terme, Telese Terme, BN
  - IRCCS "S. Maria Nascente" - Fondazione Don Gnocchi, Milan, Milan
  - IRCCS Maugeri Bari, Bari
  - Ospedale Policlinico San Martino, Genova
  - ICS Maugeri, Pavia

IPD SHARING:
Plan to Share IPD: No
A plan for wide dissemination of the results will be activated at the beginning, during and at the end of the project, through presentations at national and international conferences, and newsletters of scientific societies in the rehabilitation, neurological, and neuropsychological fields, to ensure that the results are shared with the scientific community. At the end of the project, the analysed results will be the subject of scientific publications in national and international peer-reviewed journals. The project will also be presented at regular conferences involving stakeholders (clinicians, patient and family associations) in accordance with the dissemination plan of the pnrr Fit4Med project.